CLINICAL TRIAL: NCT03827707
Title: Factors That Determine the Responses to Meal Ingestion: Effect of Ambient Noise
Brief Title: Effect of Ambient Noise on the Responses to Meal Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016H
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: meal ingestion; postprandial responses; hedonic sensations; homeostatic sensations; ambient noise
MeSH Terms: interventions — Noise; SIR1 protein, S cerevisiae

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noise (Experimental)
  Interventions: Behavioral: Noise
- Silence (Sham Comparator)
  Interventions: Behavioral: Silence

INTERVENTIONS:
Behavioral: Noise — Noise applied via headphones during 60 min after meal ingestion
  Arms: Noise
Behavioral: Silence — Headphones without sound applied during 60 min after meal ingestion
  Arms: Silence

SUMMARY:
Meal ingestion induces sensations that are influenced by a series of conditioning factors. Aim: to determine the effect of ambient noise on the sensory responses to a standard probe meal. Randomized, cross-over study in healthy subjects comparing the effect of ambient noise versus silence on the sensations induced by a probe meal. Participants (12 men) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 5 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. One study day, a noise will applied via headphones for 60 min after meal ingestion and the other day headphones without sound will applied. Perception of homeostatic sensations (hunger/ satiation, fullness) and hedonic sensations (digestive well-being, mood) will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Change in digestive well-being induced by the probe meal | 1 day
  Effect of noise on digestive well-being [measured by a 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; within subject's factors: noise and time; covariate: premeal scores).

SECONDARY OUTCOMES:
Change in fullness sensation induced by the probe meal | 1 day
  Effect of noise on fullness [measured by a 10 cm scale graded from 0 (not at all) to 10 (very much)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; within subject's factors: noise and time; covariate: premeal scores).
Change in mood induced by the probe meal | 1 day
  Effect of noise on mood [measured by a 10 cm scale graded from -5 (negative) to +5 (positive)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; within subject's factors: noise and time; covariate: premeal scores).
Change in hunger/satiety induced by the probe meal | 1 day
  Effect of noise on hunger/satiety [measured by a 10 cm scale graded from -5 (extremely hungry) to +5 (completely satiate)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; within subject's factors: noise and time; covariate: premeal scores).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Pribic T, Azpiroz F. Biogastronomy: Factors that determine the biological response to meal ingestion. Neurogastroenterol Motil. 2018 Jul;30(7):e13309. doi: 10.1111/nmo.13309. Epub 2018 Feb 2. PMID 29392797